CLINICAL TRIAL: NCT01287481
Title: Emotional Exposure and Cognitive Behavioral Therapies for Fibromyalgia
Brief Title: Pain and Stress Management for Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Michigan (Other); St. John Providence Hospital (Unknown)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AR057808 (NIH)
Record Dates: First submitted 2010-11-02; First posted 2011-02-01 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Behavioral interventions; Psychological interventions
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stress and Emotions (Experimental): Seeks to reduce stress and physical symptoms by helping individual become aware of their emotions, express them, and resolve emotional difficulties. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Stress and Emotions
- Thoughts and Behaviors (Active Comparator): Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms of fibromyalgia. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Interventions: Behavioral: Thoughts and Behaviors
- Brain and Body (Active Comparator): Seeks to help individuals improve health by educating about fibromyalgia so that one can better understand and more effectively communicate about their health. It will explain the latest scientific information about fibromyalgia, including its causes, the role of the nervous system and body, various medical and alternative treatments, and how to understand research findings.
  Interventions: Behavioral: Brain and Body

INTERVENTIONS:
Behavioral: Stress and Emotions — Focus on emotions, writing about stress, assertiveness training, role playing new ways to handle relationships, and sharing feelings and experiences with others.
  Arms: Stress and Emotions
Behavioral: Thoughts and Behaviors — Focus on cognitive and behavioral skills, such as relaxation, increasing pleasant activities, pacing, and changing ways of thinking.
  Arms: Thoughts and Behaviors
Behavioral: Brain and Body — Focus on the empowering patients by providing the latest scientific information about fibromyalgia, including causes, the role of the nervous system, and various treatments.
  Arms: Brain and Body

SUMMARY:
This interventional, randomized controlled study seeks to test the effects of an innovative emotional exposure and processing treatment that targets stress resolution, by comparing it with cognitive-behavioral therapy and a Fibromyalgia education comparison condition. The investigators also will test proposed mediators of the intervention, including improved autonomic regulation, and explore which subgroups of patients benefit the most from each approach.

ELIGIBILITY:
Inclusion Criteria:

* Meet Fibromyalgia (FM) criteria of the American College of Rheumatology (ACR)either:

  * 1990 ACR criteria including tender points
  * 2010 ACR modified clinical criteria that does not include tender points

Exclusion Criteria:

* Co-morbid autoimmune disorders, including rheumatoid arthritis and systemic lupus
* Other serious medical conditions that can impair health status independent of FM
* Current psychotic disorders (schizophrenia, bipolar disorder, etc.),dissociative identity (multiple personality) disorder, active suicide risk
* Alcohol/drug dependence in past 2 years
* Cognitive impairment or dementia
* Currently have pending (or recently received - within 2 years) FM pain related disability or workman's compensation
* Unable to fluently read or converse in English
* Planning to move from the area in the next 14 months
* Judgment of principle investigator as not appropriate for this trial or all intervention arms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment

SECONDARY OUTCOMES:
SF-12 | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
PROMIS Fatigue short form | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Pittsburgh Sleep Quality Index | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Center for Epidemiological Studies - Depression Scale | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Generalized Anxiety Disorder - 7 | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Positive and Negative Affect Schedule | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Satisfaction with Life Scale | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Multiple Ability Self-Report Questionnaire | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Patient Global Assessment of Change | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Health Care Utilization Scale | Baseline, post-treatment, 6 months post-treatment (primary endpoint), and 12 months post-treatment
Real-time Physical Activity (Actiwatch) | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Heart Rate Variability | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Levels of Emotional Awareness Scale | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Emotional Expressivity Scale | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Ambivalence over Emotional Expression | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Toronto Alexithymia Scale-20 | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Impact of Events Scale - Revised | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
BBCA - short form | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Pain Catastrophizing | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Beliefs in Pain Control Questionnaire | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Communication Thoughts and Feelings Questionnaire | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
Experimental (thumb nail pressure) threshold and tolerance ratings | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)
2010 ACR modified clinical criteria for FM, including widespread pain index | Baseline, post-treatment, and 6 months post-treatment (primary endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Lumley, Ph.D., Principal Investigator — Wayne State University
Locations (3):
- United States (3):
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - St. John Providence Hospital, Southfield, Michigan